CLINICAL TRIAL: NCT06552169
Title: The RETIRE Trial: A Randomized Phase 2 Trial of Adoptive Therapy With Treg Adoptive Cell Transfer (TRACT) To Prevent Rejection in Living Donor Kidney Transplant Recipients
Brief Title: REgulatory T Cell Therapy to Achieve Immunosuppression REduction
Acronym: RETIRE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Singulera Therapeutics Inc. (Industry)
Collaborators: Taiwan Bio Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRACT-KD-101
Record Dates: First submitted 2024-07-26; First posted 2024-08-13 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplantation
Keywords: Regulatory T cells; Treg adoptive cell transfer (TRACT); Kidney Transplantation; Graft Rejection; Autologous cell therapy; End stage renal disease; Prevention of organ transplant rejection; Tregs; Reduced immunosuppression
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — cni protein, Drosophila; Sirolimus; Everolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Standard of Care (SOC) (Active Comparator): Arm 1: SOC-Subjects randomized to Arm 1 will be followed on the prescribed 2-drug SOC immunosuppression throughout the trial.
  The study allowed SOC regimen is tacrolimus + sirolimus or everolimus.
  Interventions: Drug: Arm 1: SOC (mTOR + CNI)
- Arm 2A: TRACT/MONO mTOR (Experimental): Arm 2: TRACT/MONO- At the beginning of the trial, subjects randomized to Arm 2 will be maintained on the prescribed 2-drug SOC immunosuppression and have a single infusion of expanded Tregs (TRK-001) at Day +53 to +67 following living donor kidney transplantation.
  At Month 3 post-transplant, Arm 2 TRACT/MONO subjects will be further randomized to either Arm 2A: TRACT/MONO mTOR or Arm 2B: TRACT/MONO CNI.
  Subjects randomized to Arm 2A: TRACT/MONO mTOR who have a normal biopsy and no de novo donor specific antibodies at Month 3 will begin weaning of tacrolimus and will remain on a 1-drug regimen with either everolimus or sirolimus until the end of the trial.
  Interventions: Biological: Arm 2A: TRACT/MONO mTOR
- Arm 2B: TRACT/MONO CNI (Experimental): Arm 2: TRACT/MONO- At the beginning of the trial, subjects randomized to Arm 2 will be maintained on the prescribed 2-drug SOC immunosuppression and have a single infusion of expanded Tregs (TRK-001) at Day +53 to +67 following living donor kidney transplantation.
  At Month 3 post-transplant, Arm 2 TRACT/MONO subjects will be further randomized to either Arm 2A: TRACT/MONO mTOR or Arm 2B: TRACT/MONO CNI.
  Subjects randomized to Arm 2B: TRACT/MONO CNI who have a normal biopsy and no de novo donor specific antibodies at Month 3 will begin weaning of the mTOR medication and will remain on a 1-drug regimen with low dose tacrolimus until the end of the trial.
  Interventions: Biological: Arm 2B: TRACT/MONO CNI

INTERVENTIONS:
Drug: Arm 1: SOC (mTOR + CNI) — Subjects randomized to Arm 1 will remain on standard dual-immunosuppression therapy (CNI and mTOR) throughout the trial.
  Other Names: sirolimus or everolimus + tacrolimus
  Arms: Arm 1: Standard of Care (SOC)
Biological: Arm 2A: TRACT/MONO mTOR — All subjects will be prescribed standard of care (SOC) immunosuppressive agents. Subjects randomized to Arm 2 will be maintained on the prescribed SOC immunosuppression (tacrolimus + sirolimus or everolimus) and have a single intravenous infusion of autologous, expanded Tregs (TRK-001) at Day +53 to +67 post-transplant. At Month 3 post-transplant, Arm 2 subjects will be further randomized to receive either:
  * Arm 2A: mTOR monotherapy or
  * Arm 2B: CNI monotherapy.
  These subjects will transition to the assigned 1-drug immunosuppression regimen beginning at Month 3 post-transplant. Weaning must be completed by 12 months post-transplant.
  Subjects in Arm 2 will undergo leukapheresis to collect peripheral blood mononuclear cells required for the cellular product.
  Other Names: TRK-001 + sirolimus or everolimus
  Arms: Arm 2A: TRACT/MONO mTOR
Biological: Arm 2B: TRACT/MONO CNI — All subjects will be prescribed standard of care (SOC) immunosuppressive agents. Subjects randomized to Arm 2 will be maintained on the prescribed SOC immunosuppression (tacrolimus + sirolimus or everolimus) and have a single intravenous infusion of autologous, expanded Tregs (TRK-001) at Day +53 to +67 post-transplant. At Month 3 post-transplant, Arm 2 subjects will be further randomized to receive either:
  * Arm 2A: mTOR monotherapy or
  * Arm 2B: CNI monotherapy.
  These subjects will transition to the assigned 1-drug immunosuppression regimen beginning at Month 3 post-transplant. Weaning must be completed by 12 months post-transplant.
  Subjects in Arm 2 will undergo leukapheresis to collect peripheral blood mononuclear cells required for the cellular product.
  Other Names: TRK-001 + tacrolimus
  Arms: Arm 2B: TRACT/MONO CNI

SUMMARY:
The goal of this multi-national, multi-center, open-label, randomized Phase 2 trial is to determine the safety and efficacy of administering expanded regulatory T cells (TRK-001) to prevent allograft rejection in living donor renal transplant recipients.

Enrolled subjects will be randomized to one of 2 study arms:

Arm 1 subjects will receive standard of care immunosuppression

Arm 2 subjects will receive initial standard of care (SOC) immunosuppression and a single infusion of TRK-001. Three months after the transplant, Arm 2 subjects may be able to begin reducing their immunosuppression medication to a 1-drug regimen.

The primary outcome measures of trial are to evaluate several components indicating immunologic problems with the transplanted organ at 1-year post-transplant and to evaluate the ability for the study subjects given TRK-001 to wean to a 1-drug immunosuppression regimen.

All enrolled subjects will be followed for 5 years post-transplant.

DETAILED DESCRIPTION:
This is a prospective, multi-national, multi-center, open-label, randomized Phase 2 trial to determine the safety and efficacy of administering autologous expanded regulatory T cells (TRK-001) to prevent allograft rejection in living donor renal transplant recipients.

All subjects will be followed for 5 years post-transplant, comprising of a 2-year post-transplant follow-up period and a 3-year surveillance period.

Subjects with end-stage renal disease undergoing a living donor kidney transplant will be enrolled into the trial as follows:

Arm 1 SOC: Standard of care immunosuppression (N=14)

Arm 2 TRACT/MONO: TRK-001 and initial SOC immunosuppression weaned to monotherapy (N=20)

At Month 3 post-transplant, Arm 2 subjects will be further randomized prior to weaning to either mTOR or CNI monotherapy as follows:

Arm 2A: TRACT/MONO mTOR (N=10) or Arm 2B: TRACT/MONO CNI (N=10)

ELIGIBILITY:
Inclusion Criteria

1. Males or females aged 18-65 years as of the date of informed consent who will undergo a single organ, living donor kidney transplant.
2. Donor aged 18-65 years as of the date of organ donation. A certain degree of HLA matching between the donor and the recipient is not required.
3. Blood type compatibility between recipient and donor must be established as follows.

   Recipient A to Donor A or O; Recipient B to Donor B or O; Recipient AB to Donor A, B, AB, or O; Recipient O to Donor O.
4. No prior organ transplant of any kind.
5. Women of childbearing potential must agree to use a medically acceptable method of contraception throughout the trial. A list of the medically acceptable methods of contraception are listed in the informed consent document.
6. Male patients must agree to use birth control following the initiation of standard-of-care immunosuppression and for a minimum of 6 months following kidney transplant.
7. Subjects (recipients) must be able to understand the consent form and give written informed consent prior to any trial procedure.
8. If donor informed consent is required by IRB/IEC, donor must be able to understand the consent form and give written informed consent prior to any trial procedure. Note: Donor informed consent is required for donors participating in the research assay collections.

Exclusion Criteria Based on SOC Pre-Transplant Evaluation

1. Known sensitivity or contraindication to thymoglobulin, everolimus, sirolimus, or tacrolimus or other immunosuppression medication prescribed.
2. Subjects with an active infection considered clinically significant by an investigator that has not resolved prior to transplant.
3. Subjects with a positive flow cytometric crossmatch using donor lymphocytes and recipient serum.
4. Subjects with PRA >80% per SOC pre-transplant assessment. PRA must be repeated prior to transplant if patient receives a blood product transfusion after the initial assessment.
5. Subjects with current or historic donor specific antibodies.
6. Body Mass Index (BMI) of < 16 kg/m2 or > 38 kg/m2 per SOC pre-transplant evaluation.
7. Subjects who are pregnant or nursing mothers.
8. Subjects whose life expectancy is severely limited by diseases other than renal disease, per judgement of an investigator.
9. Ongoing active drug or alcohol substance abuse, per judgement of an investigator.
10. Major ongoing psychiatric illness or recent history of noncompliance with current medical therapy, per judgement of an investigator.
11. Significant cardiovascular disease (e.g.):

    * Significant non-correctable coronary artery disease, per judgement of an investigator
    * Ejection fraction below 30% per SOC echocardiogram if an echocardiogram is performed for an individual subject as part of their pre-transplant evaluation
    * History of recent (< 12 months) myocardial infarction at time of informed consent
    * History of recent (within 3 months) vascular intervention(s) for coronary artery disease at the time of informed consent
    * Documented arrhythmias that require a pacemaker or medical therapy for control.
12. Subjects who require use of chronic anticoagulation medications. Use of anti-platelet medications will be allowed in absence of a documented arrhythmia.
13. Malignancy within 3 years, excluding non-melanoma skin cancers such as basal cell carcinoma and squamous cell carcinoma.
14. Serologic evidence of active infection with HCV, HIV or HBV per SOC pre-transplant evaluation.
15. Subjects with a total white blood cell count < 4,000/mm3; platelet count < 50,000/mm3; triglyceride > 400 mg/dL; total cholesterol > 300 mg/dL, prothrombin time <8.4 seconds or >15.7 seconds, activated partial thromboplastin time <21.6 seconds or >42.3 seconds, fibrinogen <177 mg/dL or >598 mg/dL, and INR <0.64 or >1.4.
16. Subjects with underlying renal disease etiologies with high risk of disease recurrence such as primary focal segmental glomerulosclerosis and others per investigator discretion.
17. Subjects requiring the use of chronic immunosuppressive medication to control an underlying renal disease, or a disease with extrarenal manifestations (i.e., inflammatory bowel disease). Subjects requiring chronic or intermittent use of inhaled corticosteroids for respiratory conditions will be allowed.
18. Diabetic subjects with an HbA1c of >8%.

Exclusion Criteria Prior to Leukapheresis (Arm 2)

1. Subjects with an active infection considered clinically significant by an investigator that has not resolved prior to leukapheresis.
2. Subjects with PRA >80%, if repeated after SOC pre-transplant assessment. (PRA must be repeated prior to leukapheresis if patient receives a blood product transfusion after the initial assessment).
3. Subjects who are pregnant or nursing.
4. Subjects who received an investigational drug within 30 days prior to leukapheresis.
5. Subjects who received anti-T cell therapy within 30 days prior to leukapheresis.
6. Subjects who do not meet pre-leukapheresis clearance parameters per institutional practices or per investigator discretion.

Exclusion Criteria Prior to TRACT Cellular Product Infusion (Arm 2)

1. Subjects with an active infection considered clinically significant by the investigator that has not resolved prior to planned Treg infusion.
2. Subjects with a new, clinically significant medical condition that, per investigator opinion, would impact the ability to safely administer TRK-001.
3. Subjects who experience a rejection episode of the kidney graft prior to the planned Treg infusion.
4. Subjects who are pregnant or nursing. Women who are of childbearing potential must have a negative urine or serum pregnancy test before infusion of TRK-001.
5. Subjects who received an investigational drug within 30 days prior to infusion.
6. Subjects who received anti-T cell therapy within 30 days prior to infusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Development of de novo donor-specific antibodies | Month 12 Post-transplant
  A primary outcome measure for this study is to evaluate a composite endpoint of immunologic events against the allograft, where a failure is defined as patient-experienced immunologic events including the development of de novo donor-specific antibodies.
Biopsy-proven acute rejection | Month 12 Post-transplant
  A primary outcome measure for this study is to evaluate a composite endpoint of immunologic events against the allograft, where a failure is defined as patient-experienced immunologic events including biopsy-proven acute rejection.
Biopsy-proven subclinical rejection | Month 12 Post-transplant
  A primary outcome measure for this study is to evaluate a composite endpoint of immunologic events against the allograft, where a failure is defined as patient-experienced immunologic events including biopsy-proven subclinical rejection.
Development of significant (2+) interstitial fibrosis/tubular atrophy | Month 12 Post-transplant
  A primary outcome measure for this study is to evaluate a composite endpoint of immunologic events against the allograft, where a failure is defined as patient-experienced immunologic events including the development of significant (2+) interstitial fibrosis/tubular atrophy.
Successful taper to monotherapy (Arm 2) | Month 12 Post-transplant
  A primary outcome measure for this study is to evaluate the ability for Arm 2 subjects to successfully taper to monotherapy by one-year post-transplant.

SECONDARY OUTCOMES:
Successful maintenance of monotherapy (Arm 2) | Month 24 Post-transplant
  A secondary outcome measure for this study is to evaluate the ability for Arm 2 subjects to successfully maintain monotherapy through two-years post-transplant.
Development of de novo donor-specific antibodies | To Month 60 Post-transplant
  A secondary outcome measure for this study is to evaluate overall and composite component-specific time to immunologic failure where a failure is defined as patient-experienced immunologic events including the development of de novo donor-specific antibodies.
Biopsy-proven acute rejection | To Month 60 Post-transplant
  A secondary outcome measure for this study is to evaluate overall and composite component-specific time to immunologic failure where a failure is defined as patient-experienced immunologic events including biopsy-proven acute rejection.
Biopsy-proven subclinical rejection | To Month 60 Post-transplant
  A secondary outcome measure for this study is to evaluate overall and composite component-specific time to immunologic failure where a failure is defined as patient-experienced immunologic events including biopsy-proven subclinical rejection.
Development of significant (2+) interstitial fibrosis/tubular atrophy | To Month 60 Post-transplant
  A secondary outcome measure for this study is to evaluate overall and composite component-specific time to immunologic failure where a failure is defined as patient-experienced immunologic events including the development of significant (2+) interstitial fibrosis/tubular atrophy.
Graft loss | To Month 60 Post-transplant
  A secondary outcome measure for the study is the incidence and timing of clinical outcomes, including graft loss. Graft loss is defined as 56 consecutive days of hemodialysis or re-transplantation.
Malignancy | To Month 60 Post-transplant
  A secondary outcome measure for the study is the incidence and timing of clinical outcomes, including malignancy.
Infections | To Month 60 Post-transplant
  A secondary outcome measure for the study is the incidence and timing of clinical outcomes, including infections (bacterial, viral, fungal).
Metabolic anomalies | To Month 60 Post-transplant
  A secondary outcome measure for the study is the incidence and timing of clinical outcomes, including metabolic anomalies (e.g., diabetes mellitus, metabolic syndrome, hyperthyroidism, hypothyroidism).
Biopsy-proven acute rejection | To Month 24 Post-transplant
  A secondary outcome measure for the study is to evaluate the incidence and timing of a composite endpoint of immunologic events against the allograft, where a failure is defined as patient-experienced immunologic event, including biopsy-proven acute rejection.
Graft loss | To Month 24 Post-transplant
  A secondary outcome measure for the study is to evaluate the incidence and timing of a composite endpoint of immunologic events against the allograft, where a failure is defined as patient-experienced immunologic event, including graft loss. Graft loss is defined as 56 consecutive days of hemodialysis or re-transplantation.
Death (all cause) | To Month 24 Post-transplant
  A secondary outcome measure for the study is to evaluate the incidence and timing of a composite endpoint of immunologic events against the allograft, where a failure is defined as patient- experienced immunologic event, including all cause death.
Quality of Life Measures by using KDQOL-SF | To Month 60 Post-transplant
  The KDQOL-SF is an assessment tool designed for individuals with kidney disease to measure the impact of kidney disease and its treatment on a patient's quality of life.
Quality of Life Measures by using EQ-5D-5L | To Month 60 Post-transplant
  The EQ-5D-5L is a standardized measurement tool to evaluate health status. The questionnaire has a descriptive section and a visual analog scale.
Safety- Adverse Events | To Month 60 Post-transplant
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (4):
- Northwestern Memorial Hospital, Chicago, Illinois, United States
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Undecided